CLINICAL TRIAL: NCT00149279
Title: Randomized Controlled Trial to Evaluate Para-aortic Lymphadenectomy for Gastric Cancer (JCOG9501)
Brief Title: A Trial to Evaluate Para-aortic Lymphadenectomy for Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG9501; C000000121
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Gastric Neoplasm
Keywords: stomach neoplasms; lymph node excision; abdominal aorta
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Surgery: D2 dissection
Procedure: Surgery: D2+paraaortic dissection

SUMMARY:
To evaluate the survival benefit of para-aortic lymphadenectomy in potentially curative gastrectomy

DETAILED DESCRIPTION:
Radical gastrectomy with regional lymphadenectomy is the only curative treatment option for gastric cancer. The extent of lymphadenectomy, however, is controversial. The two European randomized trials only reported an increase in operative morbidity and mortality, but failed to show survival benefit, in the D2 lymphadenectomy group. We conducted a randomized controlled trial to compare the Japanese standard D2 and D2 + para-aortic nodal dissection.

ELIGIBILITY:
Inclusion Criteria:

- Preoperatively,

1. histologically proven adenocarcinoma
2. 75 years old or younger
3. forced expiratory volume in one second ≥ 50 %
4. arterial oxygen pressure in room air ≥ 70 mmHg
5. creatinine clearance ≥ 50 ml/min
6. written consent. Intraoperatively
7. Macroscopic T staging is T2-subserosa, T3, or T4
8. potentially curative operation is possible
9. no gross metastasis in para-aortic nodes (frozen section diagnosis not allowed)
10. peritoneal lavage cytology is negative for cancer cells

Exclusion Criteria:

1. Carcinoma in the remnant stomach
2. Borrmann type 4 (linitis plastica)
3. synchronous or metachronous malignancy in other organs except for cervical carcinoma in situ and colorectal focal cancer in adenoma
4. past history of myocardial infarction or positive results of exercise ECG
5. liver cirrhosis, or chronic liver disease with indocyanine green test ≥10%

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 520
Dates: Start 1995-07; Study Completion 2006-04

PRIMARY OUTCOMES:
overall survival

SECONDARY OUTCOMES:
relapse-free survival
operative morbidity and mortality
length of postoperative hospital stay
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuru Sasako, MD, Study Chair — Gastric Surgery Division, National Cancer Center Hospital
Locations (1):
- National Cancer Center Hospital, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Background] Sano T, Sasako M, Yamamoto S, Nashimoto A, Kurita A, Hiratsuka M, Tsujinaka T, Kinoshita T, Arai K, Yamamura Y, Okajima K. Gastric cancer surgery: morbidity and mortality results from a prospective randomized controlled trial comparing D2 and extended para-aortic lymphadenectomy--Japan Clinical Oncology Group study 9501. J Clin Oncol. 2004 Jul 15;22(14):2767-73. doi: 10.1200/JCO.2004.10.184. Epub 2004 Jun 15. PMID 15199090
- [Derived] Kurokawa Y, Sasako M, Sano T, Shibata T, Ito S, Nashimoto A, Kurita A, Kinoshita T; Japan Clinical Oncology Group. Functional outcomes after extended surgery for gastric cancer. Br J Surg. 2011 Feb;98(2):239-45. doi: 10.1002/bjs.7297. PMID 21104822
- [Derived] Sasako M, Sano T, Yamamoto S, Kurokawa Y, Nashimoto A, Kurita A, Hiratsuka M, Tsujinaka T, Kinoshita T, Arai K, Yamamura Y, Okajima K; Japan Clinical Oncology Group. D2 lymphadenectomy alone or with para-aortic nodal dissection for gastric cancer. N Engl J Med. 2008 Jul 31;359(5):453-62. doi: 10.1056/NEJMoa0707035. PMID 18669424
- See also: Related Info — http://www.jcog.jp/